CLINICAL TRIAL: NCT04059874
Title: To Assess the Safety and Efficacy of Third-line and Above Therapy of Patients With Local Advanced or Metastatic NSCLC With Combined Treatment With Launched Recombinant Humanized Anti-PD-1 Monoclonal Antibody and Donafenib Tosilate
Brief Title: Treatment of Non-small Cell Lung Cancer With PD-1 Monoclonal Antibody Combined With Donafenib Toluene Sulfonate
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhou Jianying, Chief physician, First Affiliated Hospital of Zhejiang University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZGDLH001
Record Dates: First submitted 2019-08-05; First posted 2019-08-16 (Actual); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — donafenib

STUDY DESIGN:
Intervention Model Description: This is a single-center, open, single-arm, exploratory phase Ib trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- donafenib tablets 1 (Experimental): This is the dose group was given once a day. donafenib tablets 1 100mg qd dose group
  Interventions: Drug: donafenib tablets
- donafenib tablets 2 (Experimental): This is the dose group was given twice a day. donafenib tablets 2 100mg bid dose group
  Interventions: Drug: donafenib tablets

INTERVENTIONS:
Drug: donafenib tablets — donafenib tablets 100mg qd dose group and donafenib tablets 100mg bid dose group

SUMMARY:
To assess the safety and efficacy of third-line and above therapy of patients with local advanced or metastatic non-small cell lung cancer (NSCLC) with combined treatment with launched recombinant humanized anti-PD-1 monoclonal antibody and Donafenib Tosilate

DETAILED DESCRIPTION:
Donafenib has a multi-target and dual anti-tumor effect, similar to sorafenib toluene sulfonate, and its effect is similar to that of sorafenib toluene sulfonate. Donafenib has the potential to be effective in the treatment of cancer, including advanced non-small cell lung cancer. PD-1 inhibitor has become a new therapy for advanced non-small cell lung cancer because of its strong specificity, definite efficacy, small side effects and long time of tumor control.

This is a single-center, open, single-arm, exploratory phase Ib trial. There were two dosages of donafenib (100mg qd and 100mg bid, respectively). Three to six subjects were enrolled in the dosages of 100mg qd. The investigators determined that the dosages of 100mg bid were well tolerated

ELIGIBILITY:
Inclusion Criteria:

1、18 years age or older ,male or female

2、Histologically or cytologically confirmed diagnosis of local advanced or metastatic NSCLC

3、Previously received with two or more systemic Antitumor treatments (Chemotherapy or targeted therapy). Chemotherapy treatments must include a two-drug regimen containing platinum, patients with EGFR TKI drug resistance and unknow T790M mutation, after AZD9291 treatment patients with T790M mutation could be enrolled

4、At least one measurable lesion as defined by RECIST 1.1. A previously irradiated site lesion may only be counted as a target lesion if there is clear sign of progression since the irradiation

5、Asymptomatic patients with uncontrolled brain metastases or brain metastases involving the pia mater

6、Patients must have recovered from all toxicities related to prior anticancer therapies to ≤ 2 (CTCAE v5.0). AE of Neurology must be ≤ 1

7、Life expectancy ≥ 12 weeks

8、ECOG performance status 0-1

Exclusion Criteria:

1. Small cell lung cancer (including small lung cancer mixed with non-small cell lung cancer)
2. Patients at risk of bleeding treated with antiangiogenic drugs
3. Subjects who are using immunosuppressive agents, or systemic, or absorbable topical hormone therapy for immunosuppressive purposes (dose >10mg/ dprednisone or other therapeutic hormones) and who continue to use it for 2 weeks prior to enrollment
4. Patients with active, known or suspected autoimmune diseases, including tuberculosis, HIV infection, active hepatitis, etc.
5. Patients with previous and current objective evidence of pulmonary fibrosis, interstitial pneumonia, pneumoconiosis, radioactive pneumonia, drug-related pneumonia, severe impairment of lung function, etc
6. Women who are pregnant or lactating, or who are unwilling to use contraception during the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
safety assessments | From signing ICF to 30 days after the end of treatment
  safety assessments

SECONDARY OUTCOMES:
Effective evaluation | Continue treatment until the end of treatment，an average of 12 months
  progression-free survival (PFS)
Overall response rate | Continue treatment until the end of treatment，an average of 12 months
Disease control rate | Continue treatment until the end of treatment，an average of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianying Zhou, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- The First Affiliated Hospital of College of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
No plan to share date of the trial